CLINICAL TRIAL: NCT01472133
Title: Validation of Respiration Rate Algorithms
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Engineering and Physical Sciences Research Council, UK (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Richard Beale, Clinical Director, Guy's and St Thomas' NHS Foundation Trust
Other Study IDs: 11/LO/1667
Record Dates: First submitted 2011-10-20; First posted 2011-11-16 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Respiratory Rate; Pulse Oximetry
Keywords: Respiration Rate; ECG; Pulse oximetry; Photoplethysmograph; PPG; Physiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Young Healthy Volunteers: Healthy volunteers under the age of 40
  Interventions: Other: Recording of 12 lead ECG; Other: Recording of lying and standing blood pressure; Other: Recording of chest wall movement; Other: Recording of heart rate variability; Other: Recording of ECG and Pulse oximeter waveform at rest; Other: Recording of ECG and Pulse oximeter waveform during exercise
- Older healthy volunteers: Healthy volunteers over the age of 70
  Interventions: Other: Recording of 12 lead ECG; Other: Recording of lying and standing blood pressure; Other: Recording of chest wall movement; Other: Recording of heart rate variability; Other: Recording of ECG and Pulse oximeter waveform at rest
- Patients with atrial fibrillation: Patients with permanent AF
  Interventions: Other: Recording of 12 lead ECG; Other: Recording of lying and standing blood pressure; Other: Recording of chest wall movement; Other: Recording of heart rate variability; Other: Recording of ECG and Pulse oximeter waveform at rest
- Patients with a pacemaker: Patients who have an implanted pacemaker that is continually pacing
  Interventions: Other: Recording of 12 lead ECG; Other: Recording of lying and standing blood pressure; Other: Recording of chest wall movement; Other: Recording of heart rate variability; Other: Recording of ECG and Pulse oximeter waveform at rest
- Patients with restricted chest movement: Patients whose chest expansion is less than 2.5cm
  Interventions: Other: Recording of 12 lead ECG; Other: Recording of lying and standing blood pressure; Other: Recording of heart rate variability; Other: Recording of ECG and Pulse oximeter waveform at rest

INTERVENTIONS:
Other: Recording of 12 lead ECG — Recording of 12 lead ECG
Other: Recording of lying and standing blood pressure — Recording of lying and standing blood pressure
Other: Recording of chest wall movement — Recording of chest wall movement
  Groups: Older healthy volunteers; Patients with a pacemaker; Patients with atrial fibrillation; Young Healthy Volunteers
Other: Recording of heart rate variability — Done during deep breathing and a valsalva manoeuvre
Other: Recording of ECG and Pulse oximeter waveform at rest — For 10 mins
Other: Recording of ECG and Pulse oximeter waveform during exercise — Recording of ECG and Pulse oximeter waveform during exercise
  Groups: Young Healthy Volunteers

SUMMARY:
Continuous accurate unobtrusive respiratory rate monitoring may lead to improved patient outcomes, as respiratory rate is thought to be a sensitive marker of patient deterioration. Currently systems are not suitable for long term monitoring, particularly in ambulant patients as they are too restrictive. To ensure that our algorithms are suitable for use in a clinical context we need to demonstrate their performance not only in the optimal situation, healthy volunteers at rest, but also in more challenging situations such as where the person being monitored is moving and also in patients who have conditions which may affect their physiology in such a way that the accuracy of the respiration rate estimation may be affected.

No previous study has systematically tested algorithms deriving respiratory rate from either the ECG or the photoplethysmography (PPG) waveforms in a real -world setting.

The algorithms work by looking for changes in intervals between heartbeats and also changes in the sizes of the ECG and PPG waveforms, both of which may be caused by respiration. These changes tend to diminish with increasing age and also conditions which alter the chest movement and cardiac reflexes. Thus it is important to test our algorithms' accuracy in participants exhibiting these conditions. It is also important to ensure that the calculations of respiratory rate are accurate across a range of heart rates and respiratory rates. Our testing covers all these variables.

ELIGIBILITY:
Inclusion Criteria:

* Young Healthy Volunteers

  * Participant is willing and able to give informed consent for participation in the study.
  * Male or Female, aged between 18 and 40 years old.
* Older Healthy Volunteers

  * Participant is willing and able to give informed consent for participation in the study.
  * Male or Female, aged 70 years or above.
* Patients

  * Participant is willing and able to give informed consent for participation in the study.
  * Male or Female, aged 18-70 years old.
  * Participant has one of the following conditions:
  * Atrial fibrillation
  * A permanent pacemaker that is continuously active
  * Reduced chest wall movement

Exclusion Criteria:

* Young Healthy Volunteers

  * Any condition which might increase the risk of exercise testing
  * Any history of ischaemic heart disease
  * Any history of heart failure
  * Any structural heart disease (eg: valvular lesions, hypertrophic obstructive cardiomyopathy)
  * Any abnormalities on a resting ECG
  * Deep vein thrombosis diagnosed within the last 6 months or under active treatment
  * Uncontrolled hypertension (systolic blood pressure >220 mm Hg, diastolic >120 mm Hg)
  * Aortic aneurysm
  * Aortic or cardiovascular surgery within 6 months of recruitment
  * A family history of sudden cardiac death, congenital arrhythmia syndromes or cardiomyopathy
  * Autonomic dysfunction, either previously diagnosed or upon testing by the research team
  * Any condition involving the brain or spinal cord
  * Diabetes
  * Alcohol consumption > 21 units/week for women and 28 units/week for men or a history of previous alcohol dependence.
  * Acute kidney injury
  * Chronic kidney disease stage 4 or 5
  * Any condition causing hepatic dysfunction
  * Presence of a permanent pacemaker (these participants would be eligible for the pacemaker group)
  * Reduced chest wall movement (these participants would be eligible for the reduced chest movement group)
  * Any acute infection requiring antibiotic treatment within 3 months of recruitment
  * Any other surgery or illness requiring hospitalisation within 3 months of recruitment
  * Currently taking any medication with the exception of analgesics or the oral contraceptive pill.
  * Any wound or skin condition affecting the torso which may be affected by the application of adhesive ECG dots to the skin
  * Pregnancy
  * Inability to give informed consent
* Older Healthy Volunteers

  * Any diagnosed condition primarily affecting the cardiovascular or respiratory systems
  * Symptomatic autonomic dysfunction
  * Orthostatic hypotension
  * Any condition involving the brain or spinal cord
  * Diabetes
  * Alcohol consumption > 21 units/week for women and 28 units/week for men or a history of previous alcohol dependence.
  * Acute kidney injury
  * Chronic kidney disease stage 4 or 5
  * Any condition causing hepatic dysfunction
  * Presence of a permanent pacemaker
  * Chronic Obstructive Pulmonary Disease (COPD).
  * Any muscular dystrophy
  * Kyphosis
  * Scoliosis
  * Pectus excavatum
  * Any disease involving the lungs or pleura
  * Any acute infection requiring antibiotic treatment within 3 months of recruitment
  * Any other surgery or illness requiring hospitalisation within 3 months of recruitment
  * Currently taking any medication with the exception of analgesics or the oral contraceptive pill.
  * Any wound or skin condition affecting the torso which may be affected by the application of adhesive ECG dots to the skin
  * Pregnancy
  * Inability to give informed consent
* Patients

  * Any infection which would require isolation or barrier nursing according to the hospital's infection control policy
  * Any wound or skin condition affecting the torso which may be affected by the application of adhesive ECG dots to the skin
  * Requirement for any form of artificial ventilatory support, including oxygen therapy
  * More than one of the inclusion criteria. (ie: a patient may not have both atrial fibrillation and reduced chest wall movement and be eligible for this study)
  * Inability to give informed consent

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers and hospital outpatients
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The coefficient of variation for each respiration rate algorithm | 5-6 months
  The algorithms to be tested are:
  one which calculates respiration rate (RR) from ECG only, one which calculates RR from PPG only, one which calculates RR from simultaneous ECG and PPG

SECONDARY OUTCOMES:
The coefficient of variation for the respiration rate calculated from a second pulse oximeter | 5-6 months
  Participants will wear two different PPG monitors to assess whether PPG monitors from different manufacturers introduce artefactual changes to the PPG morphology

CONTACTS AND LOCATIONS:
Overall Officials: Richard Beale, MBBS, FRCA, Principal Investigator — Guy's and St Thomas' Foundation Trust
Locations (1):
- St Thomas' Hospital, London, United Kingdom